CLINICAL TRIAL: NCT04038372
Title: Hepatitis D Virus Infection Among Hepatitis B Virus Surface Antigen Positive Individuals in Upper Egypt: Prevalence and Clinical Features
Brief Title: Hepatitis D Virus Infection Among Hepatitis B Virus Surface Antigen Positive Individuals
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Dr. Nahed A. Makhlouf, Principle Investigator, Assiut University
Other Study IDs: HDVIAHBPI
Record Dates: First submitted 2019-01-13; First posted 2019-07-30 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-04

CONDITIONS: HDV Infection; HBV Infection
Keywords: HDV; HBsAg; prevalence; Upper Egypt

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Globally, about 248 million people are chronic HBV surface antigen carriers, and about 5% of them also had hepatitis delta virus (HDV) infection as well. The prevalence of HBsAg in Egypt is intermediate (2-7%) .

Hepatitis D virus (HDV) is an incomplete RNA virus that needs hepatitis B surface antigen (HBsAg) to help its replication. HDV is considered a subviral particle because it depends on HBV for its propagation. Combined HDV- HBV infection produces more severe liver affection than HBV alone.

HDV infection leads to both of acute and chronic liver illnesses. Acute HDV infection can occur at the same time with acute HBV infection (coinfection) or can be superimposed on the top of chronic HBV infection. About 20% to 30% of coinfections of HDV and HBV in humans develop fatal fulminant hepatitis versus 2% of patients with acute hepatitis B mono-infection. Worldwide, Hepatitis D virus (HDV) infection present in more than 15 million people and it is endemic in the Middle East . In Upper Egypt, data about the prevalence, clinical, laboratory and virological characters of Hepatitis D virus-infected patients is rare.

This study aims were:

1. To estimate the prevalence of hepatitis D virus infection among HBsAg positive individuals.
2. To determine the clinical, laboratory and virological characters of HDV infected patients.

ELIGIBILITY:
Inclusion Criteria:

* HBV related liver disorder, aged 18-60 years.
* HBsAg positive individuals were divided into different clinical categories according to EASL 2012 and we revised this classification according to EASL 2017. HBeAg negative chronic infection; HBeAg positive chronic infection), Acute hepatitis, Fulminant hepatitis, Chronic hepatitis (HBeAg positive and HBeAg negative), Liver cirrhosis, and Primary HCC.

Exclusion Criteria:

* Dual infection with other viruses as HCV and/or HIV, auto-immune or alcoholic hepatitis.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: This study was a hospital-based, prospective, cross-sectional analytic one. The study was carried out on 186 HBsAg positive cases who were recruited from Tropical Medicine and Gastroenterology Department, Al Rajhi Liver Hospital, Assiut University, and Sohag University Hospital during two years.The Participants accepted to participate in the study.
Sampling Method: Probability Sample
Enrollment: 186 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
To determine Anti- HDV prevalence among HBsAg positive individuals. | 2 years
  The investigators measured Anti HDV(total) in HBsAg positive cases. Qualitative anti-HDV determination is a competitive assay, based on the ELISA technique (Enzyme-LinkedImmunosorbent), using the methodology described in the man-ufacturer's protocol. ETI-AB-DELTAK-2 (P2808) (Diasorine SPA) Italy.
To determine the prevalence of hepatitis D virus active infection. | 2 years
  The investigators did qualitative measurement of HDV PCR in Anti - HDV positive cases. Real time PCR for HDV RNA was done.

CONTACTS AND LOCATIONS:
Overall Officials: Amal A Mahmoud, MD, Assistanr Professor, Study Director — Assiut University